CLINICAL TRIAL: NCT04903626
Title: A Multicenter, Single-Arm Prospective Study to Evaluate Safety and Efficacy of GLE/PIB 8-Week Treatment in Adults and Adolescents With Acute Hepatitis C Virus (HCV) Infection
Brief Title: Study to Evaluate Adverse Events and Change in Disease Activity in Adult and Adolescent Participants With Acute Hepatitis C Virus (HCV) Infection on Treatment With Oral Tablets of Glecaprevir (GLE)/Pibrentasvir (PIB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20-350; 2020-005777-27 (EudraCT Number)
Record Dates: First submitted 2021-05-24; First posted 2021-05-26 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Acute HCV Infection; HCV Genotype 1-6; Hepatitis C; Glecaprevir; Pibrentasvir; Mavyret
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Glecaprevir/Pibrentasvir (Experimental): Participants treated once daily (QD) with glecaprevir/pibrentasvir 300 mg/120 mg for 8 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir (GLE/PIB)

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir (GLE/PIB) — Oral tablets
  Other Names: ABT-493/ABT-530; Mavyret

SUMMARY:
HCV infection is a global health problem. HCV mainly affects liver cells and causes the liver to become inflamed and damaged. This study will evaluate how safe and effective glecaprevir/pibrentasvir (GLE/PIB) is in adult and adolescent participants with acute HCV infection.

GLE/PIB is an approved drug for the treatment of chronic HCV. Around 283 participants at least 12 years of age with acute HCV Infection will be enrolled in approximately 70 sites worldwide.

Participants will receive oral tablets of GLE/PIB once daily (QD) for 8 weeks and will be followed for 12 weeks after the end of treatment.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, monitoring for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of acute HCV infection prior to enrollment, defined as a physician diagnosis of acute HCV infection, quantifiable HCV ribonucleic Acid (RNA) at screening, and at least 1 of the following:

  * Negative anti-HCV antibody, HCV RNA and/or HCV core antigen followed by a positive HCV RNA or HCV core antigen all within an 8-month period prior to screening; OR
  * Negative anti-HCV antibody, HCV RNA and/or HCV core antigen followed by a positive HCV RNA or HCV core antigen all within an 11-month period prior to screening; AND risk behavior for HCV infection within 6 months prior to positive HCV RNA or HCV core antigen; OR
  * Clinical signs and symptoms compatible with acute hepatitis [alanine aminotransferase (ALT) > 5 × upper limit of normal (ULN) and/or jaundice] in the absence of a history of chronic liver disease or other cause of acute hepatitis and positive HCV RNA or HCV core antigen all within an 8-month period prior to screening; AND risk behavior for HCV infection within 6 months prior to positive HCV RNA or HCV core antigen; OR
  * Negative anti-HCV antibody with a positive HCV RNA or HCV core antigen within a 5-month period prior to screening.
* Absence of hepatocellular carcinoma (HCC), for participants with cirrhosis, or with indeterminate cirrhosis status, as indicated by a negative ultrasound, computed tomography (CT) scan or magnetic resonance imaging (MRI) within 3 months prior to screening or a negative ultrasound at screening. Participant who has a positive ultrasound result suspicious of HCC followed by a subsequent negative CT scan or MRI or biopsy result will be eligible for the study.
* Participants documented as having no cirrhosis or as having compensated cirrhosis.

Exclusion Criteria:

* Participants with prior treatment, including interferon for this HCV infection.
* History of liver decompensation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (70):
- United States (37):
  - Arizona Health Research /ID# 233558, Chandler, Arizona
  - The Institute for Liver Health /ID# 228427, Peoria, Arizona
  - Liver Wellness Center /ID# 244933, Little Rock, Arkansas
  - AHF Research Center /ID# 254795, Beverly Hills, California
  - Velocity Clinical Research Chula Vista /ID# 238352, Chula Vista, California
  - AHF Healthcare Center- Hollywood /ID# 254794, Los Angeles, California
  - TLC Clinical Research Inc /ID# 232334, Los Angeles, California
  - University of California, Davis Comprehensive Cancer Center /ID# 230814, Sacramento, California
  - Angels Clinical Research Institute /ID# 234090, Doral, Florida
  - AIDS Healthcare Foundation (AHF) - Healthcare Center - Northpoint /ID# 254814, Fort Lauderdale, Florida
  - Midway Immunology and Research Center /ID# 229194, Ft. Pierce, Florida
  - Midland Research Group, Inc /ID# 231885, Oakland Park, Florida
  - Orlando Immunology Center /ID# 229839, Orlando, Florida
  - Tampa General Hospital /ID# 228930, Tampa, Florida
  - Duplicate_Triple O Research Institute /ID# 229928, West Palm Beach, Florida
  - Florida Medical Clinic /ID# 233489, Zephyrhills, Florida
  - Emory Midtown Infectious Disease Clinic /ID# 229927, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics /ID# 226934, Iowa City, Iowa
  - Duplicate_University of Kentucky Chandler Medical Center /ID# 231588, Lexington, Kentucky
  - University of Louisville Hospital /ID# 232139, Louisville, Kentucky
  - Mercy Medical Center /ID# 226937, Baltimore, Maryland
  - Johns Hopkins Hospital /ID# 230694, Baltimore, Maryland
  - Henry Ford Hospital /ID# 226932, Detroit, Michigan
  - University of Mississippi Medical Center /ID# 232620, Jackson, Mississippi
  - Las Vegas Research Center /ID# 255631, Las Vegas, Nevada
  - North Jersey Community Research Initiative (NJCRI) /ID# 245129, Newark, New Jersey
  - Weill Cornell Medical College /ID# 230815, New York, New York
  - Coastal Research Institute, LLC /ID# 233233, Fayetteville, North Carolina
  - The Christ Hospital /ID# 231204, Cincinnati, Ohio
  - Duplicate_University Of Cincinnati Medical Center /ID# 226922, Cincinnati, Ohio
  - Cherokee Nation Outpatient Health Center /ID# 232618, Tahlequah, Oklahoma
  - Thomas Jefferson University Hospital /ID# 232624, Philadelphia, Pennsylvania
  - University Gastroenterology /ID# 233332, Providence, Rhode Island
  - Vanderbilt University Medical Center /ID# 241282, Nashville, Tennessee
  - Liver Associates of Texas, P.A /ID# 229775, Houston, Texas
  - Digestive and Liver Disease Sp /ID# 232633, Norfolk, Virginia
  - Wisconsin Medical Center /ID# 230116, Milwaukee, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital /ID# 227167, Adelaide, South Australia
  - The Alfred Hospital /ID# 227169, Melbourne, Victoria
- Austria (3):
  - Universitaetsklinikum St. Poelten /ID# 227098, Sankt Pölten, Lower Austria
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 226985, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 226938, Vienna, Vienna
- Canada (4):
  - Vancouver Infectious Diseases Centre /ID# 227125, Vancouver, British Columbia
  - CoolAid Medical Clinic /ID# 239978, Victoria, British Columbia
  - Charlton Medical Centre /ID# 228100, Hamilton, Ontario
  - Royal Victoria Hospital / McGill University Health Centre /ID# 227126, Montreal, Quebec
- France (7):
  - CHU Montpellier - Hopital Saint Eloi /ID# 229083, Montpellier, Herault
  - CH de Tourcoing /ID# 233732, Tourcoing, Nord
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 259111, Créteil, Paris
  - HCL - Hopital de la Croix-Rousse /ID# 229077, Lyon, Rhone
  - HCL - Hopital de la Croix-Rousse /ID# 259102, Lyon, Rhone
  - AP-HP - Hopital Saint-Antoine /ID# 229070, Paris
  - Hopital Beaujon /ID# 246817, Clichy, Île-de-France Region
- Germany (6):
  - Infektiologikum /ID# 226880, Frankfurt am Main, Hesse
  - Universitaetsklinikum Bonn /ID# 226764, Bonn, North Rhine-Westphalia
  - Klinikum Dortmund gGmbH /ID# 249689, Dortmund, North Rhine-Westphalia
  - zibp-Zentrum fuer Infektiologie /ID# 226765, Berlin
  - ICH Study Center GmbH & Co KG /ID# 228162, Hamburg
  - Klinikum rechts der Isar /ID# 226783, Munich
- Italy (5):
  - IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 227080, Bologna, Emilia-Romagna
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 227079, Milan, Milano
  - Azienda Ospedaliera Universitaria Federico II /ID# 227183, Naples, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 227078, Rome, Roma
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia /ID# 227081, Foggia
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol /ID# 226698, Badalona, Barcelona
  - Hospital Parc de Salut del Mar /ID# 226696, Barcelona
  - Hospital Clinic de Barcelona /ID# 226695, Barcelona
  - Centro Sanitario Sandoval /ID# 226954, Madrid
  - Hospital Universitario Infanta Leonor /ID# 251780, Madrid
  - Duplicate_Hospital General Universitario de Valencia /ID# 226709, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Llibre JM, Boesecke C, Moon J, Lank PM, Miller MG, Fredrick LM, Welhaven A, Semizarov D, Marcinak J, Gentile I, Reiberger T, Puoti M. A single-arm phase IIIb study of 8-week glecaprevir/pibrentasvir treatment in adults with acute hepatitis C. J Hepatol. 2025 Nov 24:S0168-8278(25)02625-X. doi: 10.1016/j.jhep.2025.11.009. Online ahead of print. PMID 41297677
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glecaprevir/Pibrentasvir
Started | 286
Completed | 278
Not Completed | 8
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 1
Not completed — Other, Not Specified | 1

BASELINE CHARACTERISTICS:
Groups:
- Glecaprevir/Pibrentasvir: Participants treated QD with glecaprevir/pibrentasvir 300 mg/120 mg for 8 weeks.
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76
  Not Hispanic or Latino | 210
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 246
  Black or African American | 30
  Asian | 7
  Multiple | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in the Intention-to-Treat (ITT) Population
Description: SVR12 is defined as the hepatitis C virus (HCV) ribonucleic acid (RNA) level less than the lower limit of quantification (< LLOQ) 12 weeks after the last dose of study treatment. Efficacy was demonstrated if the lower bound of the 2-sided 95% CI for the percentage of participants achieving SVR12 was greater than 90.5%.
Time Frame: 12 weeks after last dose of study treatment (Week 20)
Population: ITT Population: all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 286
percentage of participants | 96.2 [93.2 to 97.8]

2. Secondary Outcome: Percentage of Participants Achieving SVR12 in the Modified ITT-Virologic Failure (mITT-VF) Population
Description: SVR12 is defined as the HCV RNA level < LLOQ 12 weeks after the last dose of study treatment. Efficacy was demonstrated if the lower bound of the 2-sided 95% CI for the percentage of participants achieving SVR12 was greater than 92.7%. This efficacy analysis was performed only if success was demonstrated for the primary efficacy analysis, following a fixed-sequence testing procedure.
Time Frame: 12 weeks after last dose of study treatment (Week 20)
Population: mITT-VF population: all enrolled participants who received at least one dose of study treatment, excluding those who did not achieve SVR12 for reasons other than virologic failure (i.e., those with HCV reinfection, those who did not achieve SVR12 due to early premature discontinuation of study treatment, and those who were missing HCV RNA data in the SVR12 window after backward imputation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 275
percentage of participants | 100 [98.6 to 100.0]

3. Secondary Outcome: Percentage of Participants With On-Treatment Virologic Failure in the ITT Population
Description: On-treatment virologic failure is defined as confirmed increase in HCV RNA of > 1 log^10 IU/mL above the lowest post-baseline value during treatment, confirmed HCV RNA >= 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA >= LLOQ at the end of treatment (EOT) with at least 6 weeks of treatment.
Time Frame: Up to Week 8
Population: ITT Population: all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 286
percentage of participants | 0 [0.0 to 1.3]

4. Secondary Outcome: Percentage of Participants With Post-Treatment (PT) Relapse in the ITT Population
Description: PT relapse is defined as confirmed HCV RNA >= LLOQ between the EOT and 12 weeks after the last dose of study treatment among participants who completed treatment as planned (study treatment duration >= 52 days) with HCV RNA < LLOQ at the EOT and with at least 1 PT HCV RNA value, excluding cases of reinfection.
Time Frame: Up to 12 weeks after the last dose of study treatment (Week 20)
Population: ITT Population: all enrolled participants who received at least 1 dose of study treatment. Participants who completed treatment as planned with HCV RNA < LLOQ at the EOT and with at least 1 PT HCV RNA value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 278
percentage of participants | 0 [0.0 to 1.4]

5. Secondary Outcome: Percentage of Participants With PT Reinfection With HCV in the ITT Population
Description: PT reinfection is defined as confirmed HCV RNA >= LLOQ in the PT period in a participant who had HCV RNA < LLOQ at the final treatment visit, along with the PT detection of a different HCV genotype, subtype, or clade compared with baseline.
Time Frame: Up to 12 weeks after the last dose of study treatment (Week 20)
Population: ITT Population: all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 286
percentage of participants | 0.7 [0.2 to 2.5]

ADVERSE EVENTS:
Time Frame: Screening (Day -30) through Post-treatment Week 12 (Week 20) or premature discontinuation.
Arm/Group | Glecaprevir/Pibrentasvir
All-Cause Mortality (participants affected / at risk) | 0/286
Serious Adverse Events (participants affected / at risk) | 12/286
Other Adverse Events (participants affected / at risk) | 49/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=286)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1)
RECTAL PERFORATION (Gastrointestinal disorders) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 2 (2)
BACTERAEMIA (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
MONKEYPOX (Infections and infestations) | 1 (1)
PERIORBITAL CELLULITIS (Infections and infestations) | 1 (1)
SEPTIC EMBOLUS (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CRANIOFACIAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
DRUG ABUSE (Psychiatric disorders) | 1 (1)
SUBSTANCE-INDUCED PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=286)
DIARRHOEA (Gastrointestinal disorders) | 18 (18)
FATIGUE (General disorders) | 19 (19)
NASOPHARYNGITIS (Infections and infestations) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT04903626/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT04903626/SAP_001.pdf